CLINICAL TRIAL: NCT05528315
Title: A Phase 1 Double-Blind, Randomized, Placebo-Controlled, Single and Multiple Ascending Dose Study of the Safety, Pharmacokinetics, and Pharmacodynamics of ABX-002 in Healthy Adult Subjects
Brief Title: SAD/MAD of ABX-002-1902 Investigating the Safety, Pharmacokinetics/Pharmacodynamics of in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Autobahn Therapeutics, Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ABX-002-1902
Record Dates: First submitted 2022-08-19; First posted 2022-09-06 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: MDD

STUDY DESIGN:
Intervention Model Description: Double-Blind, Randomized, Placebo-Controlled Single and Multiple Ascending Doses in Healthy Adult Subjects
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo matches appearance of ABX-002
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Single dose, ABX-002 (Experimental): Single Dose (solution) dose escalating
  Interventions: Drug: ABX-002; Drug: Placebo
- Multiple dose, ABX-002 (Experimental): Multiple Dose (solution) dose escalating
  Interventions: Drug: ABX-002; Drug: Placebo
- Formulation Comparison Solution or Capsule (Experimental): ABX-002 Single Dose TBD - Solution ABX-002 Single Dose TBD - Capsule
  Interventions: Drug: ABX-002

INTERVENTIONS:
Drug: ABX-002 — ABX-002
  Other Names: Methyl amide prodrug
Drug: Placebo — Placebo
  Arms: Multiple dose, ABX-002; Single dose, ABX-002

SUMMARY:
The study will evaluate safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single-ascending doses (SAD) and multiple ascending doses (MAD) of ABX-002 in healthy volunteers (HV)

DETAILED DESCRIPTION:
The study will evaluate safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single-ascending doses (SAD) and multiple ascending doses (MAD) of ABX-002 in healthy volunteers (HV) to identify repeated dose levels that are safe and well-tolerated.

ELIGIBILITY:
Inclusion Criteria:

* In good health, based on medical history, physical examination (including neurological examination), vital sign measurements, and laboratory safety tests
* Body mass index (BMI) 18-32 kg/m2 (inclusive)
* No clinically significant abnormality on ECG
* Must be a nonsmoker or a social smoker
* In agreement to eat a protocol-specified meal
* Women of childbearing potential (WOCBP) must have a negative urine pregnancy test at the time of the Screening Visit and before the first administration of the study drug
* WOCBP and all male subjects who are sexually active must practice effective contraception during the study and be willing and able to continue contraception for at least 90 days after their last dose of study treatment

Exclusion Criteria:

* History of any illness that, in the opinion of the study Investigator, might confound the results of the study or pose an additional risk to the subject by virtue of their participation in the study
* Mentally or legally incapacitated, has significant emotional problems
* Historical risk of suicide or according to the Investigator's clinical judgement, has made a suicide attempt in the previous 6 months, or has a history of deliberate self-harm in the past 6 months
* History of clinically significant endocrine, psychiatric, gastrointestinal, cardiovascular, peripheral vascular, neurological, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases in medical history or upon physical examination.
* History of known pre-existing liver disorders (eg, nonalcoholic fatty liver disease) and unstable liver disease History of clinically significant neoplastic disease, with the exception of adequately treated localized or in situ nonmelanoma carcinoma of the skin (ie, basal cell carcinoma) or of the cervix
* History or evidence of any of the following: myocardial infarction; cardiac valvulopathy; cardiac surgery revascularization (coronary artery bypass grafting or percutaneous transluminal coronary angioplasty); unstable angina; cerebrovascular accident, stroke, or transient ischemic attack; pacemaker; atrial fibrillation, flutter, or nonsustained or sustained ventricular tachycardia (VT); pulmonary arterial hypertension; sick sinus syndrome, second- or third-degree atrioventricular (AV) block; uncontrolled hypertension; congestive heart failure; personal or family history of sudden death or long QT syndrome; unexplained syncope or syncope within the last 3 years regardless of etiology; or history of hypokalemia
* Mean systolic blood pressure (BP) > 140 mm Hg or mean diastolic BP > 90 mm Hg
* History of multiple significant allergies and/or severe allergies (eg, food, drug, latex allergy) or has had an anaphylactic reaction or significant intolerability to prescription drugs, nonprescription drugs, or food
* Major surgery or an invasive procedure performed ≤ 3 months prior to the Screening Visit. Has donated or lost 1 unit (approximately 500 mL) of blood ≤ 56 days prior to the Screening Visit or intends to donate blood or blood products during the course of the study
* Recently received an influenza or Coronavirus Disease 2019 (COVID-19) vaccination < 1 week prior to Day -2 or intends to have an influenza or COVID-19 vaccination during the course of the study
* Subjects who are pregnant or breastfeeding
* Personal history of epilepsy or familial history of epilepsy as documented by medical records or by the history provided to the Investigator by the subject
* History of febrile seizures or seizures related to medication, intoxication, or withdrawal
* History of cataract of the lens as documented by medical records or by the history provided to the Investigator by the subject
* History of neurological abnormalities such as brain injury including traumatic injury, perinatal cerebropathy and postnatal brain damage, blood brain barrier abnormality, or cavernous angioma

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ABX-002 in healthy subjects as assessed by incidence of treatment-emergent AEs (TEAEs) and SAEs | Change from baseline
  Safety will be assessed by AEs, laboratory assessments (eg, hematology, coagulation, blood chemistry, THA markers, bone turnover biomarkers, cardiac and muscle markers, SHBG), urinalysis, pregnancy tests, vital signs (supine, orthostatic), analysis of safety ECGs, incidence and duration of selected cardiac rhythms on Holter monitoring, presence of drug-related excessive slowing or EA on EEG, slit lamp examination of the lens for cataract, and physical and neurological examinations

SECONDARY OUTCOMES:
Pharmacokinetics of ABX-002 in health subjects as assessed by maximum plasma concentration (Cmax) towards determination of the optimal PK dose | Day 1 to Day 5
  Determination of maximum plasma concentration (Cmax)
Pharmacokinetics of ABX-002 in health subjects as assessed by time to maximum concentration (Tmax) towards determination of the optimal PK dose | Day 1 to Day 5
  Determination of time to maximum concentration
Pharmacokinetics of ABX-002 in health subjects as assessed in healthy subjects as assessed by plasma exposure (AUC0-t, AUC0-inf) determination of the optimal pharmacokinetic dose | Day 1 to Day 5
  Determination of plasma exposure (AUC0-t, AUC0-inf)
Pharmacokinetics of ABX-002 in healthy subjects as assessed by terminal elimination half life (t1/2) determination of the optimal pharmacokinetic dose | Day 1 to Day 5
  Determination of terminal half life

CONTACTS AND LOCATIONS:
Overall Officials: Gudarz Davar, MD, Study Chair — Autobahn Therapeutics, Inc.
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia